CLINICAL TRIAL: NCT01806311
Title: An Open-label, Multiple-dose, Two-arm, One-sequence, Crossover Study to Evaluate the Safety and Pharmacokinetics After Oral Concurrent Administration of amlodipine10mg and candesartan32mg in Healthy Male Volunteers
Brief Title: Safety and Pharmacokinetics Study of amlodipine10mg and candesartan32mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HanAll BioPharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HAMCAO12I_1
Record Dates: First submitted 2013-03-04; First posted 2013-03-07 (Estimated); Last update posted 2025-04-20 (Actual); Status verified 2014-02

CONDITIONS: Hypertension
Keywords: Pharmacokinetics; Safety; Male
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PartA: Candesartan, Candesartan + Amolodipine (Active Comparator): Candesartan : multiple dose 32mg administered orally Amlodipine : multiple dose 10mg administered orally
  Interventions: Drug: Candesartan32mg; Drug: Amlodipine10mg
- PartB: Amlodipine, Amlodipine+Candesartan (Active Comparator): Candesartan : multiple dose 32mg administered orally Amlodipine : multiple dose 10mg administered orally
  Interventions: Drug: Candesartan32mg; Drug: Amlodipine10mg

INTERVENTIONS:
Drug: Candesartan32mg
Drug: Amlodipine10mg

SUMMARY:
Clinical trial to evalate the pharmacokinetic interactions and safety between single dose of amlodipine10mg and candesartan32mg and combiation dose amlodipine10mg with candesartan32mg in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male, Age 20 to 45
2. Subject must be willing and able to provide written informed consent to the study.

Exclusion Criteria:

1. History of any significant sickness, liver system, gall bladder system, kidney, nerve system, respiratory system, blood tumor, endocrine system, urinary system, mental disease, muscloskeletal system, immunity system, the ear, nose and throat system and cardiovascular system.
2. History of any significant gastrointestinal system and surgery of gastrointestinal.
3. History of any significant hypersensitivity to amlodipine, candesartan, aspirin, antibiotic.
4. Over 10 tobaccos a day.
5. Other condition which in the opinion of the investigator preclude endrollment into the study.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2012-12; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Part A : AUC, Cmax of Candesartan | Over a 24-hour sampling period
Par B : AUC, Cmax of Amlodipine | Over a 24-hour sampling period

SECONDARY OUTCOMES:
PartA: Cmin, tmax, CL/F of Candesartan | Over a 24-hour sampling period
PartB: Cmin, tmax, CL/F of Amlodipine | Over a 24-hour sampling period

CONTACTS AND LOCATIONS:
Overall Officials: Jang Hee Hong, Associate Professor, Principal Investigator — Chungnam national university hospital, Clinical trial center
Locations (1):
- Chungnam national university hospital,clinical trial center, Daejeon, Chungcheongbul-do, South Korea